CLINICAL TRIAL: NCT05455762
Title: Evaluating the Efficacy of Eight-week Combined Aerobic and Resistance Exercise on Clinical and Laboratory Findings and Quality of Life in Patients With Inflammatory Bowel Disease: A Randomised Controlled Trial
Brief Title: The Efficacy of Exercise Therapy in Patients With Inflammatory Bowel Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mohammad Javaherian, Dr. Mohammad Javaherian, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9511215137
Record Dates: First submitted 2022-07-10; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Inflammatory Bowel Diseases; Sarcopenia
Keywords: inflammatory bowel disease; aerobic exercise; resistance exercise; sarcopenia; quality of life
MeSH Terms: conditions — Inflammatory Bowel Diseases; Sarcopenia | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): patients in this group will participate in an 8 week program of exercise. The exercise program includes both aerobic and resistance exercise. The patients will exercise 6 days a week,3 days aerobic exercise and 3 days resistance ones. The aerobic exercise consists of 20 minutes walking. Patients will walk slowly in the first five minutes to warm up, then they walk faster and with the intensity prescribed by the physiotherapist. In the last 5 minutes the patient will walk like the first 5 minutes. The middle 10 minutes may be increased or not based on patients' weekly self-report. The resistance training include hip abduction, shoulder abduction, bridging, elbow flexion and knee extension. each of these exercises is done in 3 set of 10 repetition with one minute break between each set. Based on patients' weekly report a 0.5 kilogram weight might be added.
  Interventions: Other: Exercise
- Control group (No Intervention): The patients in this group will continue their routine life and treatment prescribed by the gastroenterologist for their condition

INTERVENTIONS:
Other: Exercise — The intervention consists of 8 week of combined resistance and aerobic exercise. Patients will exercise 6 days a week;3 days aerobic ones and 3 days resistance ones. The aerobic exercise include 20 minutes of walking divided into three parts. In the first five minute the patients walks slowly to warm up, in the next 10 minutes the patient will speedup to reach the intensity described by the physiotherapist. In the last 5 minutes the patient walks like the first five minutes. The middle 10 minutes may be increased or not based on patient's weekly report. The resistance training consists of 5 exercise; hip abduction, shoulder abduction, bridging, elbow flexion and knee extension. each of these exercises is done in 3 set of 10 repetition with one minute break between each set. Based on patients' weekly report a 0.5 kilogram weight might be added.
  Arms: Exercise group

SUMMARY:
this study aims to determine the effect of 8 weeks of exercise on the quality of life and muscle strength of patients with IBD. Patients will be randomized into 1) Intervention group: doing aerobic and resistance exercise according to physiotherapist prescription and 2) Control group: usual medical care. Both groups will continue their medications prescribed by the Gastroenterologist. After 8 weeks patients come back to the hospital for reevaluation of measured indices. The primary outcome of this study is the patient quality of life assessed by the IBDQ questionnaire. Other outcomes that will be evaluated before and after 8 weeks are muscle strength measured by a dynamometer and laboratory markers such as ESR and CRP and tool calprotectin. Also, disease activity using partial mayo score and Harvey Bradshaw score will be calculated and compared before and after treatment.

DETAILED DESCRIPTION:
Inflammatory bowel disease has a huge burden both on patients and on the health system due to its chronic nature. Studies have shown a higher prevalence of sarcopenia, a condition in which muscle mass and strength decreases, in patients with IBD compared to age and sex-matched healthy individuals. Patients with IBD are physically less active than the normal population according to a couple of researches. There has been a growing interest to evaluate the effect of exercise on the quality of life and disease severity of IBD patients in recent years.

This study aims to determine the effectiveness of combined aerobic and resistance exercise on quality of life, physical function, muscle strength, disease activity, and laboratory markers in patients with established IBD.

The researchers will invite 56 patients to the Imam Khomeini hospital complex, Tehran, Iran. All patients will be enrolled after taking informed consent. Interventions will be conducted with the coordination of the patient's physician. Patients will be randomized to the intervention or control group. Outcome measurements will be evaluated immediately before and after the interventions (8 weeks period)

ELIGIBILITY:
Inclusion Criteria:

1. Patients with IBD (UC or Chron's) confirmed by colonoscopy and pathology
2. Be able to read and write in Farsi
3. Be able to participate to exercise therapy program.

Exclusion Criteria:

1. Patients with PSC
2. Patients with cirrhosis
3. Patients with colon cancer
4. Patients on corticosteroid treatment
5. Patients' dissatisfaction to continue the study for any reason
6. Patients who exercise on a daily routine (more than 30 minutes per day)
7. Patients having any contraindication for exercise training.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life | Baseline
  assessed by IBDQ-9 questionnaire
Health-related quality of life | day 56
  assessed by IBDQ-9 questionnaire

SECONDARY OUTCOMES:
6 minute walk test | Baseline
  distance walked in 6 minute with max speed
6 minute walk test | day 56
  distance walked in 6 minute with max speed
Knee extensor muscle strength | Baseline
  muscle force measured by manual dynamometer
Knee extensor muscle strength | Day 56
  Knee extensor muscle strength
Elbow flexor muscle strength | Baseline
  muscle force measured by manual dynamometer
Elbow flexor muscle strength | Day 56
  muscle force measured by manual dynamometer
Hip flexor muscle strength | Baseline
  Muscle force measured by manual dynamometer
Hip flexor muscle strength | Day 56
  Muscle force measured by manual dynamometer
shoulder abductor muscle strength | Baseline
  Muscle force measured by manual dynamometer
shoulder abductor muscle strength | Day 56
  Muscle force measured by manual dynamometer
hand grip strength | Baseline
  Muscle force measured by manual dynamometer
hand grip strength | Day 56
  Muscle force measured by manual dynamometer
partial mayo score | Baseline
  calculated based on patient answers
partial mayo score | Day 56
  calculated based on patient answers
Harvey Bradshaw index | Baseline
  calculated based on patient answers
Harvey Bradshaw index | Day 56
  calculated based on patient answers
erythrocyte sedimentation rate | Baseline
  Measured using laboratory techniques
erythrocyte sedimentation rate | Day 56
  Measured using laboratory techniques
C-reactive protein | Baseline
  Measured using laboratory techniques
C-reactive protein | Day 56
  Measured using laboratory techniques
Stool calprotectin | Baseline
  Measured using laboratory techniques
Stool calprotectin | Day 56
  Measured using laboratory techniques

CONTACTS AND LOCATIONS:
Overall Officials: Foroogh Alborzi, M.D., Study Chair — Tehran University of Medical Sciences, Imam Khomeini hospital complex; Saeed Mirmoosavi, M.D. Student, Principal Investigator — Tehran University of Medical Sciences; Mohammad Javaherian, Ph.D., Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Imam Khomeini Hospital Complex, Tehran, Iran